CLINICAL TRIAL: NCT00766779
Title: Randomized Phase III Study Comparing Conventional Chemotherapy to Low Dose Total Body Irradiation-Based Conditioning and HCT From Related and Unrelated Donors as Consolidation Therapy for Older Patients With AML in 1st Complete Remission
Brief Title: HCT Versus CT in Elderly AML
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recommendation of DMC
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Collaborators: Acute Leukemia French Association (Other); Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); French Innovative Leukemia Organisation (Other); HOVON - Dutch Haemato-Oncology Association (Other); East German Study Group of Hematology and Oncology (OSHO) (Unknown); Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003514-34; EBMT-ALWP01/2008
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: hematopoietic cell transplantation; Acute Myeloid Leukemia; first Complete Remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transplant Arm (Experimental): Hematopoietic cell transplantation after Reduced Intensity Conditioning
  Interventions: Procedure: hematopoietic cell transplantation
- Conventional Chemotherapy (Active Comparator): The non-transplant treatment approach for consolidation
  Interventions: Drug: Non-Transplant treatment approach for consolidation

INTERVENTIONS:
Procedure: hematopoietic cell transplantation — low dose total body irradiation-based conditioning and hematopoietic cell transplantation from related and unrelated donors
  Arms: Transplant Arm
Drug: Non-Transplant treatment approach for consolidation — Patients will receive the treatment that would be otherwise applied at the local institution. The consolidation or maintenance therapy is according to the study group protocol.
  Arms: Conventional Chemotherapy

SUMMARY:
A study comparing conventional chemotherapy to low dose total body irradiation-based conditioning and hematopoietic cell transplantation from related and unrelated donors as consolidation therapy for older Patients with AML in first Complete Remission.

DETAILED DESCRIPTION:
The majority of patients with acute myelogenous leukaemia (AML) enter complete remission following induction therapy, but relapse despite consolidation and maintenance therapy. In response, post-remission treatment has been progressively intensified and results improved either by high-dose post-remission therapy with autologous hematopoietic cell transplantation (HCT) or by allogeneic HCT, which has the highest curative potential for patients with AML. Given the toxicity of dose intensification and of allogeneic HCT, however, only younger patients profit from this treatment approach

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60years and ≤ 75 years
* primary or secondary AML as defined by WHO or refractory anemia with excess of blasts (RAEB)
* First complete remission following one or two cycles of induction chemotherapy
* Chemotherapy was administered according to current participating cooperative group protocols
* Karnofsky score ≥ 70
* Written informed consent

Exclusion Criteria:

* AML FAB M3
* HIV positivity
* Participation in another clinical trial without prior consent of the coordinating investigator, patients may exceptionally take part in a further study only if

  * The second study exclusively concerns induction therapy
  * Consolidation cycle one and two are given according to the accredited study group policy
  * No investigational drugs are used post registration for the HCT vs CT in eldery AML study.
  * Documentation for the HCT vs CT in eldery AML study is not compromised. Second hand data from foreign study is not accepted

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
To evaluate Leukaemia Free Survival (LFS) after allo HCT in AML/RAEB in complete remission using matched or unrelated donors in comparison to conventional chemotherapy | 5 years

SECONDARY OUTCOMES:
To evaluate overall survival, relapse, Treatment Related Mortality (TRM) and complications after HCT | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Dietger Niederwieser, Prof, Study Chair — EBMT and OSHO; Bob Löwenberg, Prof, Study Chair — Stichting Hemato-Oncologie voor Volwassenen Nederland
Locations (48):
- The Alfred Hospital, Melbourne Victoria, Australia
- Austria (2):
  - Hanusch Krankenhaus der Wiener Gebietskrankenkasse, Vienna
  - Medizinische Universität Wien, Vienna
- Belgium (2):
  - ZNA Stuivenberg - Ziekenhuis Netwerk Antwerpen, Antwerp
  - UZ Gasthuisberg Leuven, Leuven
- France (12):
  - Centre Hospitalier Sud Amiens, Amiens
  - Hopital Femme Enfant Hématologie, Caen
  - Hôpital d'instruction des armées Percy, Clamart
  - Centre hospitalier et universitaire (CHU) d´ Estaing, Clermont-Ferrand
  - Centre hospitalier et universitaire (CHU) de Limoges, Limoges
  - Institut Paoli-Calmettes, Marseille
  - CHU de Nantes, Hôtel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre hospitalier et universitaire (CHU) de Nice, Nice
  - Hopital Saint Antoine, Paris 12ème
  - CHU du Haut Lévêque, Pessac
  - Centre Hospitalier (CH) Saint Quentin, Saint-Quentin
- Germany (17):
  - University Aachen, Aachen
  - II. Medizinische Klinik, Hämatologie/Internistische Onkologie, Augsburg
  - Charité - Campus Benjamin Franklin, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Dresden, Dresden
  - Klinik für Innere Medizin C, Greifswald
  - University of Heidelberg, Heidelberg
  - Friedrich-Schiller-Universität Jena, Jena
  - University Hospital, Leipzig
  - Universitätsklinikum Magdeburg AöR / Otto-von-Guericke Universität, Magdeburg
  - University of Münster, Münster
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - University Regensburg, Regensburg
  - Universität Rostock, Rostock
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universität Tübingen, Tübingen
  - Allogeneic Stem Cell Transplant Cente, Würzburg
- Netherlands (7):
  - Academisch Ziekenhuis bij de Universiteit Amsterdam, Amsterdam
  - VU University Medical Center Amsterdam, Amsterdam
  - University Medical Centre Groningen, Groningen
  - University Hospital Maastricht, Maastricht
  - Erasmus MC-Daniel den Hoed Cancer Centre, Rotterdam
  - University Medical Centre Utrecht, Utrecht
  - Isala klinieken, Zwolle
- Switzerland (7):
  - Kantonsspital Aarau, Aarau
  - University Hospital, Basel
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - CHUV Lausanne, Lausanne
  - Kantonsspital Luzern, Lucerne
  - University Hospital Zürich, Zurich